CLINICAL TRIAL: NCT01090921
Title: Phase II Study to Evaluate Efficacy and Safety of Single Weekly Administration of Bortezomib in Newly Diagnosed Multiple Myeloma
Brief Title: Safety and Efficacy Study of Single Weekly Bortezomib in Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Nikhil Munshi, M.D., Principal Invesetigator -- Coordinating Site, Boston VA Research Institute, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05153
Record Dates: First submitted 2010-03-15; First posted 2010-03-23 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Newly diagnosed; Newly diagnosed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Arm (Experimental): Bortezomib is administered at a dose of 1.6mg/m2 IV push over 3 to 5 seconds. Treatment is administered once a week for four weeks followed by one week off. This 5 week period is considered a treatment cycle. Dexamethasone is also administered at a dose of 40mg daily on day of and day after each dose of Bortezomib, with a dose reduction to 20mg on the same schedule if the patient cannot tolerate the higher dose of dexamethasone. The study duration for a given subject will be approximately 30 weeks.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered at a dose of 1.6 mg/m2 IV push. Treatment will be administered once a week for four weeks followed by one week off. This 5 week period is considered a treatment cycle.
  Dexamethasone will also be administered at a dose of 40mg on the day of and day after each dose of bortezomib, with a dose reduction to 20mg on the same schedule if the patient cannot tolerate the higher dose of dexamethasone.
  Other Names: Velcade

SUMMARY:
This is a research study to see if a new drug called bortezomib is useful to treat multiple myeloma in people who are newly diagnosed, and have not yet received treatment for their disease. VELCADE® (bortezomib) for Injection is a drug under development by Millennium Pharmaceuticals, Inc.

DETAILED DESCRIPTION:
This study is a multi-site study which will enroll up to 50 patients with multiple myeloma who have not had prior treatment.

Prior to starting treatment individuals will be evaluated to determine if they are eligible to participate in the study. There are certain prestudy test that are required: physical exam, blood tests, ECG, chest x-ray, skeletal survey, bone marrow aspirate and biopsy to confirm the diagnosis of multiple myeloma and to determine baseline health status.

Before beginning each treatment cycle and at the end of the study, patients will have protein studies (including blood and urine) to see if they are responding to the treatment. Before each weekly treatment cycle patients will also have blood tests for red and white blood cells and platelets, and blood chemistry tests for electrolytes, kidney and liver function, calcium and blood sugar.

Patients may receive up to 6 cycles of treatment. At the end of the study, individuals who have responded to treatment will be seen every two months to check for disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of multiple myeloma based on standard criteria.
2. Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of > 1Gm/dL and/or urine monoclonal immunoglobulin spike of > 200mg/24 hours.
3. Non-secretors must have measurable protein by Freelite or measurable disease such as plasmacytoma to be eligible.
4. Patient must not have been previously treated with chemotherapy. Prior treatment of hypercalcemia with corticosteroids, or bisphosphonates does not disqualify the patient.
5. Patient must be ineligible for autologous stem cell transplant due to one or more of the following reasons:

   * Age>65
   * Impaired renal function (creatinine≥2.0 mg/dL)
   * Impaired pulmonary function (DLCO≤50%)
   * Poor performance status (KPS≤80)
   * Other prohibitive comorbid disorder

     * 5b. Patients≥60 who decline autologous stem cell transplant are eligible for this study.
     * 5c. Patients who are eligible but wish to postpone autologous stem cell transplant are eligible for this study.
6. Karnofsky performance status>50
7. Patients treated with local radiotherapy with or without a brief exposure to steroids are eligible. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed, followed by a four week wash out period Spot RT to ≤3 vertebrae acceptable prior to entry.
8. Meets the following pretreatment laboratory criteria at Baseline (Within 14 days prior to study drug administration):

   1. Platelet count>50x10^9/L or, if the bone marrow is extensively infiltrated,>30x10^9/L
   2. Hemoglobin>8.0G/dL
   3. Absolute neutrophil count >1.0x10^9/L or, if the bone marrow is extensively infiltrated, >0.5x10^9/L
9. Meets the following pretreatment laboratory criteria for liver function tests at the screening visit conducted within 14 days of registration

   1. AST (SGOT): <3 times the upper limit of institutional laboratory normal
   2. ALT (SGPT): <3 times the upper limit of institutional laboratory normal
   3. Total bilirubin: <2 times the upper limit of institutional laboratory normal, unless clearly related to the disease
10. Women with child-bearing potential should be practicing an adequate form of contraception, as judged by the investigator (i.e. birth control pills, double barrier method, abstinence, etc.) or be surgically sterile or 12 months post-menopausal. Male subject agrees to use an acceptable method for contraception for the duration of the study.
11. Age 18 years or older
12. Has given voluntary written informed consent.

Exclusion Criteria:

1. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
2. Plasma cell leukemia
3. Impaired kidney function requiring dialysis, patients on hemodialysis are excluded
4. Receiving steroids >the equivalent of 10mg prednisone daily for other medical conditions, e.g., asthma, systemic lupus erythematosis, rheumatoid arthritis
5. Infection not controlled by antibiotics
6. HIV infection. Patients should provide consent for HIV testing according to the institution's standard practice
7. Known active hepatitis B or C
8. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix D), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
9. Second malignancy requiring concurrent treatment
10. Other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
11. Positive pregnancy test in women of childbearing potential
12. Patient has hypersensitivity to boron or mannitol.
13. Patient has ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
14. Patient has received other investigational drugs with 14 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil C. Munshi, M.D., Principal Investigator — Boston VA Research Institute, Inc.; Saem Lee, Study Chair — Boston VA Research Institute, Inc.
Locations (11):
- United States (11):
  - Little Rock VA Medical Center, Little Rock, Arkansas
  - West Los Angeles VA Medical Center, Los Angeles, California
  - San Francisco VA Medical Center, San Francisco, California
  - Eastern Colorado Health Care System, Denver, Colorado
  - West Haven VA Medical Center, West Haven, Connecticut
  - Tampa VA Medical Center, Tampa, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - VA Boston Healthcare System, Jamaica Plain, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Pittsburgh VA Medical Center, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girnius SK, Lee S, Kambhampati S, Rose MG, Mohiuddin A, Houranieh A, Zimelman A, Grady T, Mehta P, Behler C, Hayes TG, Efebera YA, Prabhala RH, Han A, Yellapragada SV, Klein CE, Roodman GD, Lichtenstein A, Munshi NC. A Phase II trial of weekly bortezomib and dexamethasone in veterans with newly diagnosed multiple myeloma not eligible for or who deferred autologous stem cell transplantation. Br J Haematol. 2015 Apr;169(1):36-43. doi: 10.1111/bjh.13243. Epub 2015 Jan 8. PMID 25572917

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib and Dexamethasone: Bortezomib is administered at a dose of 1.6mg/m2 IV push over 3 to 5 seconds. Treatment is administered once a week for four weeks followed by one week off. This 5 week period is considered a treatment cycle. Dexamethasone is also administered at a dose of 40mg daily on day of and day after each dose of Bortezomib, with a dose reduction to 20mg on the same schedule if the patient cannot tolerate the higher dose of dexamethasone. The study duration for a given subject will be approximately 30 weeks.
  Bortezomib: Bortezomib will be administered at a dose of 1.6 mg/m2 IV push. Treatment will be administered once a week for four weeks followed by one week off. This 5 week period is considered a treatment cycle.
  Dexamethasone will also be administered at a dose of 40mg on the day of and day after each dose of bortezomib, with a dose reduction to 20mg on the same schedule if the patient cannot tolerate the higher dose of dexamethasone.
Period: Overall Study
Arm/Group | Bortezomib and Dexamethasone
Started | 50
Completed | 23
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 50
Age, Customized [Mean (Full Range); unit: years]
  Age | 70.9 [50 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants at Each Response Category (Stable Disease, Minimal Response, Partial Response, Very Good Partial Response, Near Complete Response/Complete Resonse)
Description: To evaluate the response rate for weekly administered bortezomib + dexamethasone in patients with newly diagnosed multiple myeloma who are ineligible for transplant or who are eligible but wish to postpone autologous stem cell transplant.
Time Frame: Data was collected for each subject for the duration of the participation in the study, which was an average of 4.8 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 50
Participants
  Complete Response/ near Complete Response | 6
  Very Good Partial Response | 13
  Partial Response | 15
  Minimal Response | 5
  Stable Disease | 4
  Unevaluable | 7

2. Secondary Outcome: Number of Participants With Dose Reductions in Bortezomib, Dexamethasone or Both
Description: To evaluate the toxicity (safety and tolerability) of weekly bortezomib + dexamethasone in patients with newly diagnosed multiple myeloma who are ineligible for transplant or who are eligible but wish to postpone autologous stem cell transplant.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 50
Participants
  Bortezomib reductions | 8
  Dexamethasone reductions | 14
  Bortezomib and Dexamethasone reductions | 4

ADVERSE EVENTS:
Time Frame: Data was collected for each subject for the duration of the participation in the study, which was an average of 4.8 cycles.
Arm/Group | Bortezomib and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 6/50
Serious Adverse Events (participants affected / at risk) | 28/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Dexamethasone (N=50)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting/Nausea (Gastrointestinal disorders) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Asthenia (General disorders) | 4 (4)
Hyperglycemia (Endocrine disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No